CLINICAL TRIAL: NCT00437710
Title: Cardiac Study. Cellular Cardiomyoplasty of Infarcted Failed Myocardium by Autologous Intracoronary Mononuclear Bone Marrow Cell Transplantation in Humans
Brief Title: Safety and Efficacy of Bone Marrow Cell Transplantation in Humans Myocardial Infarction
Acronym: CARDIAC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Unita Sanitaria Locale di Piacenza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/2007
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2007-02

CONDITIONS: Acute Myocardial Infarction
Keywords: bone marrow, cell transplantation, stem cells, PTCA
MeSH Terms: interventions — Cell- and Tissue-Based Therapy

INTERVENTIONS:
Procedure: cell therapy, bone marrow derived stem cell

SUMMARY:
We will study in a prospective randomised fashion 50 patients who will be treated by intracoronary transplantation of autologous, mononuclear bone marrow cells (BMCs) in addition to standard therapy after MI or standard therapy.

After standard therapy for acute MI, 10 patients were transplanted with autologous mononuclear BMCs via a balloon catheter placed into the infarct-related artery during balloon dilatation (percutaneous transluminal coronary angioplasty). Another 10 patients with acute MI were treated by standard therapy alone. After

DETAILED DESCRIPTION:
Experimental and clinical data suggest that bone marrow-derived cells may contribute to the healing of myocardial infarction (MI).

ELIGIBILITY:
Inclusion Criteria:

* Recent acute transmural anterior myocardial infarction, (in agreement with WHO)
* single left anterior descending coronary artery disease
* <72 hour from the origin of symptoms
* successful primary angioplasty of the culprit lesion

Exclusion Criteria:

* screening >72 hours after infarction,
* cardiac shock, severe comorbidity, alcohol or drug dependency
* severe comorbidity (DM,renal or liver insufficiency)
* potential child bearing woman
* inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-07; Study Completion 2007-02 (Estimated)

PRIMARY OUTCOMES:
Mortality
Mortality and Morbidity
Left ventricular function

SECONDARY OUTCOMES:
Left ventricular remodeling
Heart rate variability
Baroreflex sensitivity
Stress induced myocardial ischemia
Cell dose response

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Piepoli, MD, PhD, Principal Investigator — G. da Saliceto Hospital, Regional Health Authority
Locations (1):
- G da Saliceto Hospital, Piacenza, Italy

REFERENCES:
- See also: Azienda USL Piacenza web site — http://www.ausl.pc.it/